CLINICAL TRIAL: NCT07133126
Title: Prediction of Arterial Hypotension by HPI: a Feasibility Study in Lung Resection Surgery and During Fenestrated Aortic Stenting Under General Anesthesia
Acronym: ACUMEN
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5523
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Surgery or Aortic Vascular Surgery Patients
Keywords: Non-invasive monitoring; thoracic surgery; aortic vascular surgery; HPI system; prediction; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Monitored patients: Patient undergoing a thoracic surgery or an aortic surgery will be need to be monitored during and after surgery monitored. We need to predicts and anticipates the occurrence of intraoperative arterial hypotension episodes and enables an advanced, individualized hemodynamic monitoring strategy
  Interventions: Device: Acumen monitoring

INTERVENTIONS:
Device: Acumen monitoring — Patient undergoing a thoracic surgery or an aortic surgery will be monitored as usual using the CE marked medical device ACUMEN with the intelligent HPI system.

SUMMARY:
Background: Brief review (literature data, pathology, field of study) Thoracic lung resection surgery has specific imperatives (opening of the thorax, unipulmonary ventilation, lateral decubitus operating position) that challenge the accuracy and precision of hemodynamic monitoring tools in general [1] and of systems based on arterial pressure wave analysis in particular.

The ACUMEN ClearSight® medical device enhanced by the HPI algorithm, CE marked in 2023, was developed and marketed by Edwards LifeSciences. It has been the subject of some twenty medical scientific publications since 2018 [2,3]. It is a non-invasive, single-patient sensor-type device that predicts and anticipates the occurrence of intraoperative arterial hypotension episodes and enables an advanced, individualized hemodynamic monitoring strategy.

The prediction of intraoperative arterial hypotension by the HPI machine learning algorithm is based on the invasive or non-invasive analysis of the physiological properties of the arterial pressure wave. The device is designed to optimize blood pressure management during lung resection surgery for cancer or fenestrated thoracic aortic stenting under general anesthesia. It should also enable personalized hemodynamic optimization of vascular filling and intraoperative management of vasopressor agents in patients at cardiac risk, leading ultimately to a reduction in hospital morbidity and mortality.

Non-invasive monitoring with the ClearSight® system is used routinely in the operating room at Hôpital Louis Pradel, but without the intelligent HPI system.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at moderate or high risk (ASA score ≥ 2 and/or Lee score ≥ 2)
* scheduled for lung resection by thoracotomy or video-assisted surgery or robotic surgery or fenestrated aortic stenting

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subjects scheduled for lung resection by thoracotomy or video-assisted surgery or robotic surgery and patients proposed for fenestrated aortic stenting under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Impact of ACUMEN monitoring | During the whole surgery
  Number of episodes of intraoperative arterial hypotension.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Louis PRADEL Hospices Civils de Lyon, Bron, France, France